CLINICAL TRIAL: NCT06828263
Title: Prospective Evaluation of Imaging Response Biomarkers During [177Lu]Lu-PSMA in Metastatic Castration-resistant Prostate Cancer
Acronym: 68Ga-PSMA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Johns Hopkins University (Other); LMU Klinikum (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CEMEN 2024-06
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Metastatic Disease
Keywords: Prostate cancer metastatic disease; [177Lu]Lu-PSMA; metastatic castration-resistant prostate cancer; mCRPC; LuPSMA-SPECT/CT imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lutetium-177 (177Lu) prostate-specific membrane antigen (177Lu-PSMA) is a radiolabelled small-molecule inhibitor that binds with high affinity to PSMA and delivers β particle radiation. [177Lu]Lu-PSMA-617 (Pluvicto) was approved by the U.S. Food and Drug administration (FDA) in patients with late-stage, PSMA positive metastatic castration-resistant prostate cancer (mCRPC) based on the results from the phase 3 VISION trial [1].

Early identification of tumor progression may reduce unnecessary therapy cycles and their associated risk of adverse events as well as reducing costs and improving patient care by initiating an earlier change in treatment towards a possibly more efficacious therapy.

Response Evaluation Criteria In PSMA-imaging (RECIP) version 1.0 is an evidence-based framework to evaluate therapeutic efficacy in metastatic prostate cancer using PSMA-imaging[2,3]. Interim PSMA-PET/CT by RECIP 1.0 criteria performed at 10 weeks after two cycles of PSMA theranostics ([177Lu]Lu-PSMA- 617 or [177Lu]Lu-PSMA-I&T) is prognostic for overall survival[2]. RECIP 1.0 criteria were validated based on overall survival outcome for measuring response in metastatic prostate cancer during androgen receptor-signaling inhibitors[4], as well as in early-stage prostate cancer in patients with biochemical recurrence after initial therapy[5].

Lutetium-177 is a beta therapy that also emits 11% gamma rays, which can be utilised to derive whole-body tomographic images similar to PSMA-PET/CT. Serial Lutetium-177 PSMA-targeted single photon emission tomography/computed tomography [177Lu]Lu-PSMA-SPECT/CT henceforth referred to as LuPSMASPECT/ CT has potential as an imaging response biomarker for 177Lu-PSMA therapy. This principle enables image quantitation and evaluation after every treatment dose. SPECT/CT post [177Lu]Lu-PSMA administration represents a potentially cost-effective alternative to interim PSMA-PET/CT.

Preliminary results have shown a good correlation between changes in LuPSMASPECT/ CT during PSMA theranostics and clinical outcome. LuPSMA-SPECT/CT can provide effective response information as early as 6 weeks after initiation of [177Lu]Lu-PSMA-I&T, i.e. any increase in total tumor volume on SPECT/CT imaging was associated with shorter PSA-PFS (median: 3.7 vs 6.7 months; HR, 2.5; 95% CI 1.5-4.2; p<0.001)[6]. Changes in total tumor volume on 12-week LuPSMASPECT/ CT were also found to be correlated with progression-free survival after [177Lu]Lu-PSMA-I&T[7].

The growing evidence suggesting that LuPSMA-SPECT/CT is a new, early surrogate marker for assessing response to treatment has several potential upsides, including the potential replacement of interim PSMA-PET/CT, therefore costsaving, radiation exposure-saving, and SPECT/CT imaging being more convenient and widely available.

Given that data regarding SPECT/CT-based treatment response monitoring during PSMA theranostics are limited, this study aims to prospectively investigate the role of LuPSMA-SPECT/CT imaging for response evaluation during treatment with [177Lu]Lu-PSMA in mCRPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or older with proven adenocarcinoma of the prostate
* Diagnosis of progressive metastatic castration-resistant prostate cancer.
* Progression or intolerance on a novel anti-androgen therapy (i.e. abiraterone, enzalutamide, apalutamide or darolutamide)
* Prior therapy with at least one taxane-based chemotherapy during the course of prostate cancer or the patient is symptomatic and assessed as unfit for chemotherapy.
* ECOG Performance status 0 to 2

Exclusion Criteria:

* Patient opposed to the use of his data for clinical research.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the investigator's department only
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2043-06 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Confirm prospectively the prognostic value of post-therapy SPECT/CT imaging for response evaluation during [177Lu]Lu- PSMA | From treatment initiation to at least 12 months after treatment initiation
  Associations between response on 177Lu-PSMA-SPECT with OS, defined as the associations between best overall response achieved on LuPSMA-SPECT/CT at any time during treatment with overall survival. The associations will be considered positive if difference in OS between PD vs nPD is statistically significant (p<0.05) as per Kaplan-Meier analysis (log-rank test).

SECONDARY OUTCOMES:
Validate prognostic value of interim PSMA-PET/CT performed at 10 weeks after initiation of [177Lu]Lu-PSMA | From treatment initiation to at least 12 months after treatment initiation
  Associations between response on 10-week PSMA-PET/CT with OS. The associations will be considered positive if difference in OS between PD vs nPD or PD vs SD vs PR according to RECIP 1.0 is statistically significant (p<0.05) as per Kaplan-Meier analysis (log-rank test).
To compare cost-effectiveness of SPECT/CT versus PET/CT treatment response strategy | From treatment initiation to at least 12 months after treatment initiation
  Determine clinical significance of performing interim PSMA-PET/CT versus SPECT/CT for treatment response evaluation during [177Lu]Lu- PSMA. Percentage of participants with ≥1 new lesion detected on interim PSMA-PET that is not detected on LuPSMA-SPECT imaging performed at 6 weeks and/or 12 weeks. The interim PSMA-PET will be considered of clinical value if patients with ≥1 new lesion detected only on interim PSMAPET have statistically significant (p<0.05) shorter PFS and/or OS compared to patients without new lesions detected on PSMA-PET and/or LuPSMASPECT, as per Kaplan-Meier analysis (log-rank test).
Investigate added value of interim [18F]FDG PET to PSMA-PET/CT for response evaluation during [177Lu]Lu-PSMA | From treatment initiation to at least 12 months after treatment initiation
  Determine the added value of interim [18F]FDG-PET to PSMA-PET/CT for response evaluation during [177Lu]Lu-PSMA. Presence of new lesion, volume and tumor uptake changing on [18F]FDG-PET performed at 10 weeks. The interim FDG-PET will be considered of clinical value if patients with progression on FDG-PET have statistically significant (p<0.05) shorter PFS and OS compared to patients without new lesions detected on PSMA-PET and/or LuPSMA-SPECT and/or CT images, as per Kaplan-Meier analysis (log-rank test).
Determine clinical impact of performing interim PSMA-PET/CT versus LuPSMA-SPECT/CT for response evaluation during [177Lu]Lu-PSMA | From treatment initiation to at least 12 months after treatment initiation
  Correlations of LuPSMA-SPECT/CT progression-free survival (LuSPECTPFS) with OS. LuSPECT-PFS is defined as the time from treatment initiation to the date of progression on 177Lu-PSMA-SPECT/CT according to RECIP 1.0 criteria or death due to any cause, whichever occurs first [3].
  The correlations will be significant if the Spearman coefficient r is higher than 0.6 and p<0.01 [8].
Prognostic value of 177Lu-PSMA-SPECT/CT/PSMA PET derived tumor burden quantitative parameters for OS | From treatment initiation to at least 12 months after treatment initiation
  Prognostic value of 177Lu-PSMA-SPECT/CT/PSMA PET derived tumor burden quantitative parameters for OS. Total tumor volume, SUVmax, SUVmean and more advanced parameters obtained using artificial intelligence algorithms will be assessed. Association between algorithm predicted outcome with observed outcome will be tested
Inter-reader agreement | From treatment initiation to at least 12 months after treatment initiation
  Inter-reader agreement for response evaluation using interim LuPSMA- SPECT/CT and PSMA-PET/CT according to RECIP 1.0.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gafita A, Djaileb L, Rauscher I, Fendler WP, Hadaschik B, Rowe SP, Herrmann K, Calais J, Rettig M, Eiber M, Weber M, Benz MR, Farolfi A. Response Evaluation Criteria in PSMA PET/CT (RECIP 1.0) in Metastatic Castration-resistant Prostate Cancer. Radiology. 2023 Jul;308(1):e222148. doi: 10.1148/radiol.222148. PMID 37432081
- [Result] Pathmanandavel S, Crumbaker M, Ho B, Yam AO, Wilson P, Niman R, Ayers M, Sharma S, Hickey A, Eu P, Stockler M, Martin AJ, Joshua AM, Nguyen A, Emmett L. Evaluation of 177Lu-PSMA-617 SPECT/CT Quantitation as a Response Biomarker Within a Prospective 177Lu-PSMA-617 and NOX66 Combination Trial (LuPIN). J Nucl Med. 2023 Feb;64(2):221-226. doi: 10.2967/jnumed.122.264398. Epub 2022 Aug 25. PMID 36008120
- [Result] John N, Pathmanandavel S, Crumbaker M, Counter W, Ho B, Yam AO, Wilson P, Niman R, Ayers M, Poole A, Hickey A, Agrawal S, Perkins G, Kallinen A, Eslick E, Stockler MR, Joshua AM, Nguyen A, Emmett L. 177Lu-PSMA SPECT Quantitation at 6 Weeks (Dose 2) Predicts Short Progression-Free Survival for Patients Undergoing 177Lu-PSMA-I&T Therapy. J Nucl Med. 2023 Mar;64(3):410-415. doi: 10.2967/jnumed.122.264677. Epub 2022 Sep 8. PMID 36215568
- [Result] Kendrick J, Francis RJ, Hassan GM, Rowshanfarzad P, Ong JS, McCarthy M, Alexander S, Ebert MA. Prognostic utility of RECIP 1.0 with manual and AI-based segmentations in biochemically recurrent prostate cancer from [68Ga]Ga-PSMA-11 PET images. Eur J Nucl Med Mol Imaging. 2023 Nov;50(13):4077-4086. doi: 10.1007/s00259-023-06382-2. Epub 2023 Aug 8. PMID 37550494
- [Result] Shagera QA, Karfis I, Kristanto P, Spyridon S, Diamand R, Santapau A, Peltier A, Roumeguere T, Flamen P, Artigas C. PSMA PET/CT for Response Assessment and Overall Survival Prediction in Patients with Metastatic Castration-Resistant Prostate Cancer Treated with Androgen Receptor Pathway Inhibitors. J Nucl Med. 2023 Dec 1;64(12):1869-1875. doi: 10.2967/jnumed.123.265874. PMID 37770114
- [Result] Gafita A, Rauscher I, Weber M, Hadaschik B, Wang H, Armstrong WR, Tauber R, Grogan TR, Czernin J, Rettig MB, Herrmann K, Calais J, Weber WA, Benz MR, Fendler WP, Eiber M. Novel Framework for Treatment Response Evaluation Using PSMA PET/CT in Patients with Metastatic Castration-Resistant Prostate Cancer (RECIP 1.0): An International Multicenter Study. J Nucl Med. 2022 Nov;63(11):1651-1658. doi: 10.2967/jnumed.121.263072. Epub 2022 Apr 14. PMID 35422442
- [Result] Sartor O, de Bono J, Chi KN, Fizazi K, Herrmann K, Rahbar K, Tagawa ST, Nordquist LT, Vaishampayan N, El-Haddad G, Park CH, Beer TM, Armour A, Perez-Contreras WJ, DeSilvio M, Kpamegan E, Gericke G, Messmann RA, Morris MJ, Krause BJ; VISION Investigators. Lutetium-177-PSMA-617 for Metastatic Castration-Resistant Prostate Cancer. N Engl J Med. 2021 Sep 16;385(12):1091-1103. doi: 10.1056/NEJMoa2107322. Epub 2021 Jun 23. PMID 34161051